CLINICAL TRIAL: NCT03943134
Title: A Multicenter, Ambispective, Clinical Outcomes Registry Study of Avive® Soft Tissue Membrane Utilization in Selected Applications of Acute Trauma of the Upper Extremity
Brief Title: Registry of Avive® Soft Tissue Membrane Utilization in Selected Applications of Acute Trauma of the Upper Extremity
Acronym: ASSIST
Status: Terminated | Type: Observational
Why Stopped: Axogen suspended market availability of the Avive® Soft Tissue Membrane effective June 1, 2021. This decision was not related to any safety concerns or product quality issues.
Sponsor: Axogen Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: ASM-CP-001
Record Dates: First submitted 2019-05-06; First posted 2019-05-09 (Actual); Last update posted 2025-08-20 (Actual); Status verified 2025-08

CONDITIONS: Acute Upper Extremity Trauma
Keywords: Acute Trauma; Upper Extremity Trauma; Acute Upper Extremity Trauma; Avive; Peripheral Nerve Injury; Nerve Repair
MeSH Terms: conditions — Peripheral Nerve Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Avive® Soft Tissue Membrane: Subjects with utilization of Avive® Soft Tissue Membrane on an impacted but intact nerve during a surgical procedure for one of the following targeted acute upper extremity traumas (selected injuries): Spaghetti Wrist, Distal Radius Fracture, Medial Epicondyle Fracture, Flexor Tenolysis at Wrist, and Ballistic Injuries in the Forearm and/or Hand.
  Interventions: Other: Minimally Processed Human Umbilical Cord Membrane
- Standard Surgical Procedures - Control Arm: Subjects who have undergone surgical procedures for the same selected injuries, but without placement of a surgical implant on an impacted but intact nerve.
  Interventions: Other: Standard Surgical Procedures

INTERVENTIONS:
Other: Minimally Processed Human Umbilical Cord Membrane — Implantation of minimally processed human umbilical cord membrane at the time of surgery
  Groups: Avive® Soft Tissue Membrane
Other: Standard Surgical Procedures — Standard surgical intervention for at least one targeted acute upper extremity trauma
  Groups: Standard Surgical Procedures - Control Arm

SUMMARY:
A registry study to evaluate the role of Avive® Soft Tissue Membrane in the management of nerve injury associated with acute trauma in the upper extremity.

DETAILED DESCRIPTION:
This is a multicenter outcomes registry study of Avive® Soft Tissue Membrane in the management of nerve injuries associated with selected upper extremity acute trauma. The study will evaluate clinical condition, economic impact, and functional outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects 5 to 70 years of age, inclusive;
2. Sign and date an IRB/IEC -approved written informed consent form (ICF) prior to initiation of any study activities;

   1. Group One only: Subject enrollment (ICF completion) must be completed within 2 weeks (7-14 days) post-operatively of the targeted surgical procedure;
   2. Group Two Retrospective subjects only: Sign and date an IRB/IEC - approved written informed consent form (ICF) prior to initiation of any study activities if required per the governing IRB;
3. Group One only: Subjects who have undergone placement of Avive® Soft Tissue Membrane over at least one exposed nerve, circumferentially, or as an overlay between the exposed nerve(s) and the surrounding wound bed during surgical intervention following one or more of the following targeted acute upper extremity traumas (selected injuries): Spaghetti Wrist, Distal Radius Fractures, Medial Epicondyle Fractures, Flexor Tenolysis at Wrist, and/or Ballistic Injuries in the Forearm and/or Hand. This surgical intervention must have been completed within 60 days from the date of injury;
4. Group Two only: Subjects who have undergone surgical intervention for one or more of the following targeted acute upper extremity traumas (selected injuries): Spaghetti Wrist, Distal Radius Fractures, Medial Epicondyle Fractures, Flexor Tenolysis at Wrist, and Ballistic Injuries in the Forearm and/or Hand in the past 5 years without placement of a surgical implant over the exposed nerve, circumferentially, or as an overlay between the exposed nerve(s) and the surrounding wound bed during surgical intervention. This surgical intervention must have been completed within 60 days from the date of injury;
5. Group Two only: Subjects must have at least 1 qualifying post-operative injury assessment;
6. Subject is willing and able to comply with all aspects of the treatment and evaluation schedule.

Exclusion Criteria:

1. Subjects with complete transection of all nerves affected by one or more of the following selected injuries: Spaghetti Wrist, Distal Radius Fractures, Medial Epicondyle Fractures, Flexor Tenolysis at Wrist, and Ballistic Injuries in the Forearm and/or Hand. Subjects with nerve transection(s) must also have ≥1 affected nerve intact (non-transected) for treatment with Avive® Soft Tissue Membrane (Group One) or without treatment with a surgical implant (Group Two);
2. Subjects with Type 1 Diabetes Mellitus or Type 2 Diabetes Mellitus requiring regular insulin therapy;
3. Subjects who are currently receiving, or have previously received, treatment with chemotherapy, radiation therapy, or other known treatment which affects the growth of the neural and/or vascular system;
4. Subjects that are currently taking, or have previously used, a medication that is known to cause peripheral neuropathy;
5. Subjects with a history of chronic ischemic condition of the upper extremity; and
6. Any subject who, at the discretion of the Investigator, is not suitable for inclusion in the study.

Ages: 5 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Subjects who have had surgical intervention for one or more of the targeted acute upper extremity traumas
Sampling Method: Non-Probability Sample
Enrollment: 7 (Actual)
Dates: Start 2018-12-01 (Actual); Primary Completion 2020-12-17 (Actual); Study Completion 2020-12-17 (Actual)

PRIMARY OUTCOMES:
Changes in QuickDASH (Disabilities of Arm, Shoulder, Hand) score at 2,4,8,12,16,24, and 52 post-operative weeks (Adult subjects only). | 2, 4, 8, 12, 16, 24, and 52 weeks
  Adult patients will be assessed for changes in functional status using the QuickDASH outcomes assessment. The quickDASH is an abbreviated version of the original DASH outcomes measures and is comprised of an 11-item patient reported questionnaire used to assess physical function and severity of symptoms in patients with musculoskeletal disorders of the upper limb. Each of the items in the quickDASH use a 5-point Likert scale to assess the corresponding severity or functional parameter. The outcome measure is scored based on the formula ([sum of n responses)/n]-1)(25), where n represents the number of completed items. Computed scores range from 0 (no disability) to 100 (most severe disability).
Changes in PROMIS Pediatric Upper Extremity/Parent Proxy Upper Extremity (PUE/PPUE) outcomes assessment at 2,4,8,12,16, 24, and 52 post-operative weeks (Pediatric subjects only) | 2, 4, 8, 12, 16, 24, and 52 weeks
  The Patient Reported Outcome Measurement Information System (PROMIS®) - pediatric Related Measures is a set of person-centered measures that evaluates and monitors a patient's physical health and pain (pediatric patients). Short forms containing fixed sets of 4-10 items or questions are included for each domain. All PROMIS scores are presented as T-scores where the T-score is the standardized score with a mean of 50 (range 20-80) and a standard deviation of 10. Higher scores indicate more of the concept being measures where sometimes the concept is desirable (e.g., physical function) and sometimes this it is undesirable (e.g., fatigue). PROMIS instruments are scored using item-level calibrations based on response patterns by HealthMeasures Scoring Service (https://www.assessmentcenter.net/ac_scoringservice).
Change in Visual Analogue Scale (VAS) For Pain Score at 2, 4, 8, 12, 16, 24, and 52 post-operative weeks | 2, 4, 8, 12, 16, 24, and 52 weeks
  The Visual Analog Scale (VAS) For Pain is a patient reported outcomes scale whereby the patient indicates his/her current pain level by making a mark on a continuous horizontal 10 centimeter (100 millimeter) line. The distance from the 0 millimeter to the patient's mark corresponds to the amount of pain the subject is currently experiencing. VAS for Pain data are recorded as the number of millimeters from the left of the line to the patients mark across the range of 0-100 millimeters, with 0 millimeter representing no pain and 100 millimeters representing "the worst pain imaginable".
Changes in Reported Pain Using the Faces Pain Scale-Revised Scale (FPS-R) assessment at 2, 4, 8, 12, 16, 24, and 52 post-operative weeks | 2, 4, 8, 12, 16, 24, and 52 weeks
  Pediatric patients will be assessed for changes in patient reported outcomes using the FPS-R. The Faces Pain Scale - Revised (FPS-R) is a self-report measure of pain intensity developed for children. It was adapted from the Faces Pain Scale to make it possible to score the sensation of pain on the widelya accepted calculated 0-to-10 metric. The scale shows a close linear relationship with visual analog pain scales across the age range of 4-16 years. The calculated score ranges from 0 ("no pain") to 10 ("very much pain").
Changes in patient reported health status Using SF-36 patient reported health survey at 2, 4, 8, 12, 16, 24, and 52 post-operative weeks | 2, 4, 8, 12, 16, 24, and 52 weeks
  Adult patients will be assessed for changes in patient reported health status using the SF-36 patient reported health survey. The SF-36 measures overall health status and consists of eight scaled scores which are the weighted sums of the questions in their section. Each scale is directly translated into a 0-100 metric scale. Scoring ranges from 0 (maximum disability to 100 (no disability).
Changes in KINDL Health-Related Quality of Life questionnaire for children at 2, 4, 8, 12, 16, 24, and 52 post-operative weeks | 2, 4, 8, 12, 16, 24, and 52 weeks
  The KINDL is a generic quality of life instrument used to assess Health-Related Quality of Life in children and adolescents aged 3 years and older. The questionnaire is comprised of 24 items which assess various quality of life domains using 5-point Likert scales. Calculated scores range from 0 (lower quality of life) to 100 (higher quality of life).
Change in Patient Rated Wrist Evaluation | 2, 4, 8, 12, 16, 24, and 52 weeks
  Patients will be assessed for changes in patient reported outcomes using the Patient Rated Wrist Evaluation (PRWE)(Applicable to Injuries Affecting the Wrist)
Change in Sensory Function as measured by Medical Research Council Classification (MRCC) for Sensory Recovery | 2, 4, 8, 12, 16, 24, and 52 weeks
  Patients will be assessed for changes in 2-Point Discrimination on a scale from 0 to 4 with 0 representing no sensation and 4 representing a 2-point discrimination measure between 2-6 representing normal sensation.
Change in Motor Function as measured by Medical Research Council Classification (MRCC) for Motor Recovery | 2, 4, 8, 12, 16, 24, and 52 weeks
  Patients will be assessed for changes in muscle strength measured on a scale from 0 to 5, with 0 equal to no movement and 5 equal to normal muscle contraction against resistance.
Change in Motor Function as measured by Grip and Pinch Strength | 2, 4, 8, 12, 16, 24, and 52 weeks
  Patients will be assessed for changes in grip and pinch strength measured in kg force
Change in Motor Function as measured by Range of Motion | 2, 4, 8, 12, 16, 24, and 52 weeks
  Patients will be assessed for changes in range of motion measured in degrees
Change in Tinel's Sign | 2, 4, 8, 12, 16, 24, and 52 weeks
  Patients will be assessed for presence of Tinel's Sign
Incidence of Adverse Events Associated with the Placement of Avive Soft Tissue Membrane | 2, 4, 8, 12, 16, 24, and 52 weeks
  Adverse events are defined as any untoward event experienced by a patient that is related to the nerve repair (whether or not considered product related by the Principal Investigator or Sponsor) or any even that has changed adversely in nature, severity or frequency.
Health Care Economic Impact based on Resource Utilization and Associated Costs | 2, 4, 8, 12, 16, 24, and 52 weeks
  Patients will be assessed for cost of procedures, post-procedure medications, rehabilitation, re-hospitalization

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Florida Orthopaedic Institute, Tampa, Florida
  - Indiana Hand to Shoulder Center, Indianapolis, Indiana
  - Upstate Hand Center, Spartanburg, South Carolina

IPD SHARING:
Plan to Share IPD: No